CLINICAL TRIAL: NCT04709588
Title: Hydrolyzed Collagen Combined With Djulis and Green Caviar Improve Skin Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EWISH-20190917-01
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): subjects drank 50 ml every night for 14, 28 days
  Interventions: Dietary Supplement: placebo group
- collagen drinks (Experimental): subjects drank 50 ml every night for 14, 28 days
  Interventions: Dietary Supplement: collagen drinkss

INTERVENTIONS:
Dietary Supplement: placebo group — subjects drank 50 ml every night for 14, 28 days
  Arms: placebo group
Dietary Supplement: collagen drinkss — subjects drank 50 ml every night for 14, 28 days
  Arms: collagen drinks

SUMMARY:
Collagen combined with djulis and green caviar improve skin condition

DETAILED DESCRIPTION:
Using collagen drinks combined fish collagen with djulis, and green caviar to improve skin condition.

ELIGIBILITY:
Inclusion Criteria:

1. Dry skin
2. Rough skin
3. Large pores
4. Dark yellow complexion
5. Sagging skin

Exclusion Criteria:

1. Skin disorders
2. Liver diseases
3. Kidney diseases
4. Allergy to cosmetics, drugs, or foods
5. Pregnant and lactating women
6. People who had any cosmetic procedures before 4 weeks of the study
7. Area of facial spot over 3 cm2
8. Vegan
9. People who took collagen supplements in the past 3 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
skin moisture | subjects drank 50 ml every night for 28 days
  using corneometer CM825 to examine skin moisture (The higher the value, the more water content, C.U., corneometer units )
skin elasticity | subjects drank 50 ml every night for 28 days
  using cutometer dual MPA580 to examine skin elasticity (The closer the R2 value is to 1, the better the elasticity and no unit)
skin gloss | subjects drank 50 ml every night for 28 days
  using probe system GL2000 & MPA10 to examine skin gloss (The higher the value, the higher the gloss, no unit)
skin spot | subjects drank 50 ml every night for 28 days
  usig VISIA-CR to examine skin spot (The higher the value, the larger the pore area, mm2)
skin wrinkle | subjects drank 50 ml every night for 28 days
  using VISIOSCAN-VC20 to examine skin wrinkle (The higher the value, the more wrinkles, surface evaluation of wrinkles, SEW)
skin roughness | subjects drank 50 ml every night for 28 days
  using VISIOSCAN-VC98 to examine skin roughness (The higher the value, the higher the roughness, surface evaluation of roughness, SEr)
skin smoothness | subjects drank 50 ml every night for 28 days
  using VISIOSCAN-VC98 to examine skin smoothness (The lower the value, the higher the smoothness, surface evaluation of smoothness, SEsm)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fu Chiang, Ph.D, Principal Investigator — Research & Design Center, TCI CO., Ltd
Locations (1):
- Research & Design Center, TCI CO., Ltd, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No